CLINICAL TRIAL: NCT03818542
Title: A Phase 1b Multi-Center Pharmacodynamic Study to Assess the Effects of Multiple Study Drug Regimens in Subjects With Newly Diagnosed Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: A Study to Assess the Effects of Multiple Study Drug Regimens in Subjects With Newly Diagnosed Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M19-228
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Squamous Cell Carcinoma; Cancer; ABBV-927; ABBV-368; ABBV-181; tumor resection; immunotherapeutic drug
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Neoplasms | interventions — budigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: ABBV-181 IV (Experimental): A single dose of ABBV-181 administered via intravenous (IV) infusion on Day 1.
  Interventions: Drug: ABBV-181
- Arm 2: ABBV-368 IV (Experimental): A single dose of ABBV-368 administered via intravenous (IV) infusion on Day 1.
  Interventions: Drug: ABBV-368
- Arm 3: ABBV-927 IV (Experimental): A single dose of ABBV-927 administered via intravenous (IV) infusion on Day 1.
  Interventions: Drug: ABBV-927
- Arm 4: ABBV-927 IT (Experimental): A single dose of ABBV-927 administered via intratumoral (IT) injection on Day 1.
  Interventions: Drug: ABBV-927

INTERVENTIONS:
Drug: ABBV-181 — intravenous infusion
  Arms: Arm 1: ABBV-181 IV
Drug: ABBV-368 — intravenous infusion
  Arms: Arm 2: ABBV-368 IV
Drug: ABBV-927 — intravenous infusion
  Arms: Arm 3: ABBV-927 IV
Drug: ABBV-927 — intratumoral injection
  Arms: Arm 4: ABBV-927 IT

SUMMARY:
A study evaluating the safety, pharmacokinetics, and biomarker profiles of multiple study drugs as monotherapy in subjects with newly diagnosed, treatment-naïve locally advanced squamous cell carcinoma of the head and neck who are candidates for surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed stage 3 to 4B squamous cell carcinoma of the oral cavity, oropharynx, larynx, or hypopharynx who are candidates for surgical resection and are treatment-naïve. Participants must have been determined to be candidates for surgical resection by a multidisciplinary team including a surgeon, a medical oncologist, and a radiation oncologist.
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1 and life expectancy of more than 3 months.
* Must consent to provide the tumor tissues for analyses as described in the protocol.
* Must have adequate bone marrow function (without any growth factors or transfusions within 2 weeks prior to the first dose), kidney and liver function, with all laboratory values criteria detailed in the protocol.

Exclusion Criteria:

* Has received live vaccine within 28 days prior to the first dose of study drug.
* Has a history of inflammatory bowel disease, a history of or ongoing pneumonitis or interstitial lung disease, had major surgery ≤ 28 days prior to the first dose of study drug and the surgical wound is not fully healed.
* Participants with hypopharyngeal or laryngeal tumors will not be candidates for Arm 4 of the study (IT injection of ABBV-927).
* Requires use of an immunosuppressive medication within 14 days prior to the first dose of the study drug; exceptions are described in the protocol.
* Has a confirmed positive test results for human immunodeficiency virus, or have active hepatitis A, B or C.
* Has a history of primary immunodeficiency, allogeneic bone marrow transplantation, solid organ transplantation, or previous clinical diagnosis of tuberculosis.
* Has a history of any other malignancy within the past 3 years except for successfully treated non-melanoma skin cancer or localized carcinoma in situ that is considered cured or adequately treated by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Changes in Gene Expression | Baseline (before initiation of drug treatment) and after surgical resection (up to 120 days after study drug administration)
  The primary biomarker endpoint is to assess immune activation gene changes in the tumor microenvironment associated with T cell infiltration and activation, comparing baseline biopsy to surgical resection following drug treatment.

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of Study Drug | Up to approximately 120 days
  Maximum Serum Concentration (Cmax) of study drug
Time to Maximum Plasma Concentration (Tmax) of Study Drug | Up to approximately 120 days
  Time to Maximum Plasma Concentration (Tmax) of study drug
Area Under the Plasma Concentration-time Curve of Study Drug in Plasma | Up to approximately 120 days
  Area Under the Plasma Concentration-time Curve (AUC) of study drug in plasma

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (3):
- United States (3):
  - Massachusetts General Hospital /ID# 207392, Boston, Massachusetts
  - University of Michigan /ID# 210181, Ann Arbor, Michigan
  - MD Anderson Cancer Center /ID# 208749, Houston, Texas

IPD SHARING:
Plan to Share IPD: No